CLINICAL TRIAL: NCT03502564
Title: Co-occurring Eating Disorders and Posttraumatic Stress Disorder: Facilitating Full and Sustained Recovery Through Empirically-Based Concurrent Treatment
Brief Title: Integrated Treatment for Co-occurring Eating Disorders and Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kathryn Trottier, Staff Psychologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB# 15-8826-A
Record Dates: First submitted 2017-11-14; First posted 2018-04-18 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: PostTraumatic Stress Disorder; Eating Disorder
Keywords: Posttraumatic stress disorder; Eating disorders; Cognitive behavior therapy; Cognitive processing therapy; Randomized controlled trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT for ED only (Active Comparator): In this arm, participants will receive CBT for ED following intensive ED treatment (see intervention section for description).
  Interventions: Behavioral: CBT for ED
- Concurrent CBT for ED and PTSD (Experimental): In this arm, participants will receive concurrent CBT for ED and PTSD following intensive treatment. (see intervention section for description).
  Interventions: Behavioral: Concurrent CBT for ED and PTSD

INTERVENTIONS:
Behavioral: CBT for ED — Cognitive behavior therapy (CBT) for eating disorders (ED) is a 16-session individual therapy protocol which will focus on maintaining improvements in eating following intensive treatment, as well as addressing overconcern with weight/shape. Interventions will be adopted from the Enhanced CBT for ED manual.
  Other Names: CBT for ED only
  Arms: CBT for ED only
Behavioral: Concurrent CBT for ED and PTSD — The concurrent ED and PTSD intervention will consist of 16 sessions of CBT for both PTSD and for ED (ED interventions described above). CBT for PTSD will be based on interventions in the Cognitive Processing Therapy (CPT) manual.
  Other Names: CBT for ED and PTSD
  Arms: Concurrent CBT for ED and PTSD

SUMMARY:
Although psychotherapy for eating disorders (EDs) can be effective, approximately 50% of those who complete a course of the best available therapy continue to have significant ED symptoms at the end of treatment. Posttraumatic stress disorder (PTSD) commonly co-occurs with EDs and is thought to be one reason why some individuals do not remit from their ED with best available treatment or relapse following treatment. In particular, ED behaviours can function as coping methods for PTSD symptoms, and thus interfere with successful and lasting ED recovery. The main objective of this initial treatment trial is to determine whether a concurrent treatment approach, in which PTSD symptoms are treated at the same time as ED symptoms, provides an advantage over standard ED treatment by successfully alleviating PTSD symptoms.

Forty participants who have both an ED and PTSD will be assigned to receive either (1) standard ED psychotherapy alone or (2) standard ED psychotherapy concurrent with PTSD psychotherapy. After treatment, participants will be followed for a period of 6 months to determine whether improvements made during therapy are maintained after treatment. ED and PTSD symptoms, as well as concomitant symptoms (e.g., anxiety and depression) will be assessed immediately before and after treatment, as well as 3 and 6 months after treatment.

DETAILED DESCRIPTION:
Standard ED treatment is characterized by partial response in many individuals, and the risk of relapse is high. This, in combination with significant rates of comorbid PTSD, evidence that trauma history can negatively impact ED treatment outcome, and the observation that PTSD may be a central ED maintaining factor in these individuals, has led us to develop a program of research aimed at demonstrating that the alleviation of PTSD symptoms concurrent with ED treatment facilitates a fuller and sustained ED recovery for these individuals.

The specific aims of this initial randomized controlled trial (RCT) are to determine: (1) the immediate and short-term efficacy of concurrent evidence-based ED and PTSD treatment in reducing PTSD symptoms relative to standard ED treatment; and (2) estimates of the effect sizes of concurrent treatment on ED symptomatology relative to standard ED treatment at post-treatment and follow-up.

Primary Hypothesis:

1. Concurrent CBT for ED and PTSD will result in significantly greater improvements in clinician-rated PTSD symptoms at post-treatment, as well as at 3- and 6-month follow-up compared with CBT for ED alone.

   Secondary Hypotheses:
2. Concurrent CBT for ED and PTSD will result in significantly greater improvements in self-reported PTSD symptoms at post-treatment, as well as at 3- and 6-month follow-up compared with CBT for ED alone.
3. Concurrent CBT for ED and PTSD will result in significantly greater improvements in concomitant symptoms (e.g., anxiety and depression) at post-treatment, as well as at 3- and 6-month follow-up compared with CBT for ED alone.

Exploratory Research Questions

1. What proportion of participants experience reliable improvement in ED symptomatology and what proportion experience reliable deterioration in ED symptomatology over the course of each treatment?
2. What is the relative efficacy of concurrent CBT for ED and PTSD versus CBT for ED alone in reducing functional deficits at post-treatment, and 3- and 6-month follow-up?
3. What is the relative efficacy of concurrent CBT for ED and PTSD versus CBT for ED alone in improving other concomitant symptoms at post-treatment, and 3- and 6-month follow-up?

METHOD:

Following a course of intensive ED treatment in the inpatient or day hospital ED program at University Health Network (UHN), participants will be randomly assigned to receive either individually-administered: (1) standard CBT for ED alone or (2) concurrent CBT for ED and PTSD. Participants in both conditions will receive 16 sessions. Eleven of the 16 concurrent CBT for ED and PTSD sessions will be 90 minutes long in order to accommodate the administration of CBT for ED and PTSD. Participants in the CBT for ED alone condition will also receive eleven 90-minute sessions in order to control for time in therapy. In the CBT for ED condition, therapists will have more time to cover the ED-related content. Accordingly, both treatments will consist of eleven 90-minute sessions and five 50-minute sessions, with two sessions per week for the first 8 sessions, weekly sessions for the following 6 sessions, and biweekly for the final two sessions.

Participants will be assessed pre-CBT for ED/PTSD and post-CBT for ED/PTSD, as well as 3 and 6 months after treatment. The assessors will be blind to treatment condition, and an intent-to-treat (ITT) approach to data collection and analysis will be adopted. ED and PTSD symptoms will also be assessed on a weekly basis during the study treatments.

STATISTICS:

1. Primary hypothesis: Changes in clinician-rated PTSD symptoms will be analyzed using multilevel modeling, including a random effect for time and fixed effects for therapy condition, time, and the condition by time interaction. Change in PTSD symptoms over time and differences between the conditions over time will be examined. Empirically derived covariates that significantly reduce error variance will be used. Cohen's d effect sizes will be calculated.
2. Secondary hypotheses: Changes in self-reported PTSD symptoms, anxiety, and depresion will be analyzed using multilevel modeling, including a random effect for time and fixed effects for therapy condition, time, and the condition by time interaction. Change in PTSD symptoms, anxiety, and depression over time and differences between the conditions over time will be examined. Empirically derived covariates that significantly reduce error variance will be used. Cohen's d effect sizes will be calculated.
3. The proportion of participants who experience reliable improvement and the proportion who experience reliable deterioration in ED symptomatology in each therapy condition will be calculated using reliable change criteria (Jacobson & Truax, 1991).
4. The proportion of participants meeting diagnostic criteria for PTSD and an eating disorder will be compared between conditions at post-treatment and follow-up.
5. Changes in other concomitant symptoms and functional deficits will be analyzed using multilevel modeling as described above.

ELIGIBILITY:
Inclusion Criteria:

* have had a minimum dose of intensive eating disorder treatment in the Toronto General Hospital Eating Disorder Program, defined as 6 weeks or longer
* have current Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) diagnoses of an eating disorder and PTSD
* be on a stable (or no) psychotropic medication regimen for at least 4 weeks

Exclusion Criteria:

* current body mass index less than 18.5
* current substance use disorder involving dependence
* current psychosis
* current bipolar episode
* medical treatment or other condition known to influence eating and/or weight
* current participation in another psychosocial treatment for ED or trauma
* current participation in any treatment study for ED or trauma
* has previously received cognitive processing therapy for PTSD

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in clinician-assessed PTSD symptoms | pre-treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  Change in PTSD symptoms will be assessed using the Clinician-Administered PTSD Scale (CAPS; Weathers et al., 2013). Scores range from 0-80 with a higher score representing higher severity.

SECONDARY OUTCOMES:
Change in self-reported PTSD symptoms | pre-treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  The PTSD Checklist (PCL; Weathers, Litz, Keane, Palemeri, Marx, & Schnurr, 2013) will provide a measure of change in self-reported PTSD symptoms. Scores can range from 0-80 with a higher score indicating higher severity.
Change in anxiety | pre-treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  Change in anxiety will be assessed with the anxiety scale of the Depression Anxiety Stress Scales (DASS; Lovibond & Lovibond, 1995). Scores can range from 0-42 with a higher score reflecting higher anxiety.
Change in depression | pre-treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  Change in depression will be assessed with the depression scale of the Depression Anxiety Stress Scales (DASS; Lovibond & Lovibond, 1995). Scores can range from 0-42 with a higher score reflecting higher depression.

OTHER OUTCOMES:
Change in clinician-rated eating disorder (ED) symptomatology | pre-treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  Change in clinician-rated frequency of ED symptoms and severity of ED features will be assessed via the Eating Disorder Examination (EDE; Fairburn, Cooper, & O'Connor, 2014)
Functional deficits | pre-treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  The Social Adjustment Scale Self-Report (SASSR; Weissman & Bothwell, 1976) will provide an outcome measure of functional deficits across six primary domains: work; social and leisure activities; extended family relationships; role in spousal relationship; role in parental relationships; and role in family unit relationship. Higher scores indicate greater impairment of functioning. Scores range from 1-5.
Change in self-reported eating disorder (ED) symptomatology | pre-treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  Change in frequency of self-reported ED symptoms and severity of ED features will be assessed via the questionnaire version of the EDE (EDE-Q; Fairburn & Beglin, 2008).
Change in Beck depression scores | pre-treatment, weekly during treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  Change in depression symptoms will be assessed with the Beck Depression Inventory (BDI-II; Beck, Steer, & Brown, 1996). Scores can range from 0-63 with a higher score reflecting a higher level of depression.
Change in emotion regulation | pre-treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  Emotion regulation will be assessed with the Difficulties with Emotion Regulation Scale (DERS; Gratz & Roemer, 2004). The total score can range from 36-180, with higher scores suggesting greater emotion dysregulation. The DERS has 6 subscales.
Change in shame | pre-treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  Shame will be assessed using the Experiences of Shame Scale (ESS; Andrews, Qian, & Valentine, 2002). The total score can range from 25-100. The ESS has 3 subscales.
Change in schematic beliefs. | pre-treatment, end of treatment (after approximately 14 weeks), 3- and 6-month follow up
  Schematic beliefs will be assessed using the Young Schema Questionnaire (YSQ; Young, 1998). The YSQ has 15 subscales and scores on the subscales range from 5-30.
Treatment acceptability and satisfaction | after session 4, end of treatment (after approximately 14 weeks)
  Treatment acceptability and satisfaction will be measured with investigator constructed Likert Scales.
Weekly change in self-reported PTSD symptoms | weekly over approximately 14 weeks
  The PTSD Checklist (PCL; Weathers, Litz, Keane, Palemeri, Marx, & Schnurr, 2013) weekly version will provide a measure of change in self-reported PTSD symptoms over the course of treatment. Scores can range from 0-80 with a higher score indicating higher severity.
Behavioural urges over the course of treatment | weekly over approximately 14 weeks
  Self-reported urges for eating disorder behaviours, self-injury and substance use will be assessed using an investigator-constructed questionnaire on a weekly basis over the course of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Trottier, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Eating Disorder Program; Toronto General Hospital; University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Hamblen JL, Schnurr PP, Rosenberg A, Eftekhari A. A guide to the literature on psychotherapy for PTSD. Psychiatric Annals 39(6): 348-354, 2009.
- [Background] Watts BV, Schnurr PP, Mayo L, Young-Xu Y, Weeks WB, Friedman MJ. Meta-analysis of the efficacy of treatments for posttraumatic stress disorder. J Clin Psychiatry. 2013 Jun;74(6):e541-50. doi: 10.4088/JCP.12r08225. PMID 23842024
- [Background] Resick PA, Monson CM, Chard KM. Cognitive processing therapy: Veteran/military version. Washington, DC: Department of Veterans' Affairs. 2007 Jun.
- [Background] Weathers FW, Blake DD, Schnurr PP, Kaloupek DG, Marx BP, Keane TM. The clinician-administered PTSD scale for DSM-5 (CAPS-5). Interview available from the National Center for PTSD at www. ptsd. va. gov. 2013 Aug 6.
- [Background] Weathers FW, Litz BT, Keane TM, Palmieri PA, Marx BP, Schnurr PP. The ptsd checklist for dsm-5 (pcl-5). Scale available from the National Center for PTSD at www. ptsd. va. gov. 2013.
- [Background] Beck AT, Steer RA, Brown GK. Beck Depression Inventory. San Antonio, TX, United States: The psychological corporation.1996.
- [Background] Lovibond SH, Lovibond PF. Manual for the Depression Anxiety Stress Scales. (2nd. Ed.) Sydney: Psychology Foundation. 1995.
- [Background] Fairburn CG, Cooper Z, O'Connor M. The Eating Disorder Examination (EDE 17). Interview available from http://www.credo-oxford.com/pdfs/EDE_17.0D.pdf. 2014.
- [Background] Fairburn CG, Beglin A. Eating Disorder Examination Questionnaire (EDE-Q 6.0). In C. G. Fairburn, Cognitive Behavior Therapy and Eating Disorders (pp. 309-313). New York: Guilford. 2008.
- [Background] Weissman MM, Bothwell S. Assessment of social adjustment by patient self-report. Arch Gen Psychiatry. 1976 Sep;33(9):1111-5. doi: 10.1001/archpsyc.1976.01770090101010. PMID 962494